CLINICAL TRIAL: NCT01619176
Title: Non Inferiority Trial for the Study of Acupuncture on Rheumatoid Arthritis
Brief Title: Acupuncture Study on Rheumatoid Arthritis, Monitoring Microbiome and Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, Christine Nardini, Principal Investigator, Chinese Academy of Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: acumicro
Record Dates: First submitted 2012-06-05; First posted 2012-06-14 (Estimated); Results first posted 2023-09-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; blood; gut intestinal microbiome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Anti-Inflammatory Agents, Non-Steroidal; Leflunomide; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture plus conventional treatment (methotrexate+leflunomide+non-steroid anti-inflammatory drugs)
  Interventions: Drug: methotrexate; Drug: non-steroidal anti-inflammatory drug (NSAID); Drug: leflunomide; Procedure: Acupuncture
- Control (Active Comparator): Conventional treatment (methotrexate+leflunomide+non-steroid anti-inflammatory drugs)
  Interventions: Drug: methotrexate; Drug: non-steroidal anti-inflammatory drug (NSAID); Drug: leflunomide

INTERVENTIONS:
Drug: methotrexate — methotrexate: 7.5mg/week to 15mg/week for 3 months
  Arms: Control
Drug: non-steroidal anti-inflammatory drug (NSAID) — NSAID: 100mg twice a day for 3 months
  Arms: Control
Drug: leflunomide — leflunomide: 20mg/day for 3 months
  Arms: Control
Drug: methotrexate — methotrexate: 7.5mg/week to 15mg/week for 3 months
  Arms: Acupuncture
Drug: non-steroidal anti-inflammatory drug (NSAID) — NSAID: 100mg twice a day for 3 months
  Arms: Acupuncture
Drug: leflunomide — leflunomide: 20mg/day for 3 months
  Arms: Acupuncture
Procedure: Acupuncture — 30 minutes acupuncture every other day for 3 months.
  Basic acupoints: Zusanli, st36; Taixi，KI3）; Shenxu, BL23 Additional acupoints due to personal condition: Waiguan，SJ5; Baxie，Ex-UE9;Yinlingquan，(SP9）; Quchi，LI11; Yanglingquan，GB34; Xuehai，SP10; Dazhu，BL11; Dazhui，DU14; Pixu，BL20.
  Arms: Acupuncture

SUMMARY:
Acupuncture is used and recommended by the WHO for the treatment of Rheumatoid Arthritis.

The molecular bases of this recommendation are not known, the investigators want to compare with the usage of high-throughput molecular technologies the variations occurring in patients treated with acupuncture and conventional treatment with the ones treated with conventional treatment only. The investigators observe the variations in blood and in the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be diagnosed as the first or second stage of rheumatoid Arthritis (RA) and checked with X ray for additional diagnose.
* diagnosed for RA according to ACR(1987)
* the patient should be in the active stage of the disease, defined as：

  1. swollen joints >3
  2. tender joints > 5
  3. any one of the following： (c1.) morning stiffness lasting more than 45 minutes (c2.) Erythrocyte Sedimentation Rate (ESR) >= 28mm/h (c3.) C-reactive protein (CRP)>= 12mg/L
* Should not be resistant to MTX nor leflunomide
* Blood test should satisfy:

  1. Hemoglobin (Hb)>=85g/L
  2. White cell >=3.5 10+9/L
  3. Platelets >= 100 10+9/L
  4. Liver function: serum alanine aminotransaminase (ALT), aspartate transaminase (AST) and total bilirubin (TBil) should be less than 1.5 times the upper limit of normal (ULN)
  5. Kidney function: Serum creatinine (Cr) level should be less than ULN.
  6. Pregnancy test should be negative
* should be positive for anti-cyclic citrullinated protein antibodies (anti-CCP).
* should agree to sign the informed consent

Exclusion Criteria:

* Serious diseases affecting liver, kidney, heart and lung, or diseases related to hematologic，endocrine and nervous systems. .
* Be treated by MTX or Leflunomide in the last 3 months.
* Be treated with cortical hormone （could be intramuscular injection, intravenous injection or injection to articular cavity） in the last 4 weeks.
* Be treated with biological agents, such as antagonist of TNF-alpha,IL-6, and CD20 mono antibody in the last 3 months.
* Be treated by chronic medicine, such as immunosuppressive agent, Penicillamine, chloroquine and gold based Disease-modifying antirheumatic drugs (DMARDs) in the last 3 months.
* Pregnant and breast-feeding woman
* Having history of serious drug allergy
* In the acute or chronic phase of infection (such as lung diseases)
* Easy bleeding patients or patients with local skin infection (only for acupuncture)
* The patients cannot accept acupuncture (only for acupuncture)
* Be treated with acupuncture in the past 3 months（only for acupuncture）.
* No pregnant and breast-feeding woman.
* No history of serious drug allergy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Nardini, PhD, Study Chair — Key laboratory of Computational Biology,Chines Academy of Sciences-Max Planck Institute-CAS MPG PICB; Christine Nardini, PhD, Study Chair — Consiglio Nazionale delle Ricerche Istituto per le Applicazioni del Calcolo "Mauro Picone"; Yuanhua Liu, Principal Investigator — Shanghai Institute of Biochemistry and Cell Biology, CAS, Shanghai, PRC; Yongying Liang, Principal Investigator — Guanghua Hospital, Shanghai, PRC; Xiaoyuan Zhou, Principal Investigator — Group of Clinical Genomic Networks, Shanghai Institutes for Biological Sciences, CAS-MPG, China; Jennifer E. Dent, Principal Investigator — Group of Clinical Genomic Networks, Shanghai Institutes for Biological Sciences, CAS-MPG, China; Ting Jiang, Principal Investigator — Department of Neurology, University of California, San Francisco, USA; Ding Qin, Principal Investigator — Guanghua Hospital, Shanghai, PRC; Youtao Lu, Principal Investigator — Group of Clinical Genomic Networks, Shanghai Institutes for Biological Sciences, CAS-MPG, China; Dongyi He, Study Director — Guanghua Hospital, Shanghai, PRC
Locations (1):
- Shanghai GuangHua Hospital of integrated traditional and western medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Liu, Y. et al. (2023). Wound Healing from Bench to Bedside: A PPPM Bridge Between Physical Therapies and Chronic Inflammation. In: Podbielska, H., Kapalla, M. (eds) Predictive, Preventive, and Personalised Medicine: From Bench to Bedside. Advances in Predictive, Preventive and Personalised Medicine, vol 17. Springer, Cham. https://doi.org/10.1007/978-3-031-34884-6_12
- See also: Book chapter — https://link.springer.com/chapter/10.1007/978-3-031-34884-6_12#citeas
- Available data/document: Individual Participant Data Set: GSE59526 — http://www.ncbi.nlm.nih.gov/geo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Quality of biological sampling was not good enough to grant production of quality omic data
Groups:
- Acupuncture: Acupuncture plus conventional treatment (methotrexate+leflunomide+non-steroid anti-inflammatory drugs)
  methotrexate: methotrexate: 7.5mg/week to 15mg/week for 3 months
  non-steroidal anti-inflammatory drug (NSAID): NSAID: 100mg twice a day for 3 months
  leflunomide: leflunomide: 20mg/day for 3 months
  Acupuncture: 30 minutes acupuncture every other day for 3 months.
  Basic acupoints: Zusanli, st36; Taixi，KI3）; Shenxu, BL23 Additional acupoints due to personal condition: Waiguan，SJ5; Baxie，Ex-UE9;Yinlingquan，(SP9）; Quchi，LI11; Yanglingquan，GB34; Xuehai，SP10; Dazhu，BL11; Dazhui，DU14; Pixu，BL20.
Period: Overall Study
Arm/Group | Acupuncture | Control
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Control | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (13.08) | 48.0 (10.3) | 48.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 6 | 4 | 10
RF(IU/mL) [Mean (Standard Deviation); unit: IU/mL] — Rheumatoid Factor
  IU/mL | 246.25 (235.3) | 382.4 (409.1) | 314.3 (317.4)
CRP(mg/L) [Mean (Standard Deviation); unit: mg/L] — C-reactive protein Population: The sum does not match the total due to missing data
  mg/L
    number analyzed (Participants) | 3 | 4 | 7
    (all) | 9.8 (5.3) | 24.6 (22.3) | 18.27 (17.9)
ESR（mm/h) [Mean (Standard Deviation); unit: mm/h] — Erythrocyte Sedimentation Rate
  mm/h | 53.2 (45.5) | 71.2 (60.2) | 60.4 (49.4)
hemoglobin(g/L) [Mean (Standard Deviation); unit: g/L] | 119.5 (13.1) | 113.5 (24.1) | 117.1 (16.4)
White cell number(10^9 cells/L) [Mean (Standard Deviation); unit: 10^9 cells/L] | 6.0 (1.8) | 5.2 (3.6) | 5.7 (2.4)
neutrophile granulocyte(%) [Mean (Standard Deviation); unit: % of cells] | 61 (6.5) | 69.0 (6.1) | 64.2 (6.9)
Lymphocyte(%) [Mean (Standard Deviation); unit: % of cells] | 30.3 (6.6) | 21.0 (3.2) | 26.6 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: ACR20 Response Rate at 3 Weeks
Description: ACR criteria stands for: American College of Rheumatology Criteria. ACR criteria measures improvement in tender or swollen joint counts and improvement in three of the following five parameters:
  acute phase reactant (such as sedimentation rate) patient assessment physician assessment pain scale disability/functional questionnaire
  The number indicates the percentage of improvement in tender or swollen joint counts as well percentage improvement in three of the other five criteria (patient's assessment of pain, a physician's global assessment of disease, a patient's global assessment of disease, physical function as assessed by the Health Assessment Questionnaire-Disability Index (HAQ-DI), and the level of acute-phase reactant)
Time Frame: From baseline to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 2 | 4
Participants | 0 | 1

2. Primary Outcome: ACR20 Response Rate at 3 Months
Description: as for outcome 1
Time Frame: From baseline to three months
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 6 | 4
Participants | 5 | 3

3. Secondary Outcome: ACR50 Response Rate at 3 Weeks
Description: as for outcome 1
Time Frame: From baseline to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 2 | 4
Participants | 0 | 1

4. Secondary Outcome: ACR50 Response Rate at 3 Months
Description: as for outcome 1
Time Frame: From baseline to three months
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 6 | 4
Participants | 2 | 1

5. Secondary Outcome: ACR70 Response Rate at 3 Weeks
Description: as for outcome 1
Time Frame: From baseline to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

6. Secondary Outcome: ACR70 Response Rate at 3 Months
Description: as for outcome 1
Time Frame: From baseline to three months
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 6 | 4
Participants | 0 | 1

7. Secondary Outcome: DAS28 at Baseline
Description: The DAS28 (disease activity score) considers 28 tender and swollen joint counts, general health (GH; patient assessment of disease activity using a 100 mm visual analogue scale (VAS) with 0 = best, 100 = worst), plus levels of an acute phase reactant (either the level of erythrocyte sedimentation rate ESR (mm/h) or C-reactive protein CRP (mg/litre)). DAS28 values were calculated as follows: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96; DAS28 (ESR) = 0.56*√(TJC28)+0.28*√(SJC28)+0.014*GH+0.70*ln(ESR), where TJC = tender joint count and SJC = swollen joint count.
  The scale does not have bounds. DAS28 total score < 2,6 means remission DAS28 total score ranged between 2.6-3.2 means inactive disease; DAS28 total score ranged between 3.3-5.1 means moderate disease activity; DAS28 total score >5.1 means very active disease
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 6 | 4
units on a scale | 4.98 (1.13) | 6.8 (1.97)

8. Secondary Outcome: DAS28 at 3 Weeks
Description: The DAS28 (disease activity score) considers 28 tender and swollen joint counts, general health (GH; patient assessment of disease activity using a 100 mm visual analogue scale (VAS) with 0 = best, 100 = worst), plus levels of an acute phase reactant (either the level of erythrocyte sedimentation rate ESR (mm/h) or C-reactive protein CRP (mg/litre)). DAS28 values were calculated as follows: DAS28 (CRP) = 0.56*√(TJC28) +0.28*√(SJC28)+0.014*GH+0.36*ln(CRP+1)+0.96; DAS28 (ESR) = 0.56*√(TJC28)+0.28*√(SJC28)+0.014*GH+0.70*ln(ESR), where TJC = tender joint count and SJC = swollen joint count.
  The scale does not have bounds. DAS28 total score < 2,6 means remission DAS28 total score ranged between 0-3.2 means inactive disease; DAS28 total score ranged between 3.3-5.1 means moderate disease activity; DAS28 total score >5.1 means very active disease
Time Frame: At 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 2 | 4
units on a scale | 5 (0.14) | 5.27 (1.15)

9. Secondary Outcome: DAS28 at 3 Months
Description: as for outcome 8
Time Frame: At 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 6 | 4
units on a scale | 3.85 (0.59) | 4.5 (0.6)

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | Acupuncture | Control
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If discussion include scientific publication there is no restriction